CLINICAL TRIAL: NCT06808178
Title: The EFFECT of KINESIO TAPING and LOW LEVEL LASER THERAPY in PATIENT with POST MASTECTOMY RELATED LYMPHEDEMA on GIRTH MEASUREMENT
Brief Title: EFFECT of KINESIO TAPING and LASER THERAPY in PATIENT with LYMPHEDEMA on GIRTH MEASUREMENT
Acronym: LYMPHEDEMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Awad Ramadan Elkholy, Lecturer of physical therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/02012024/Zaki
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Lymphedema; Breast Cancer Stage II
Keywords: laser taping
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: 60 females with BCRL will be recruited in this study for 4 weeks , their age ranged from 400 to 55 years old with stege 1,2 lymphedema and randomly divided into 3 equal groups: 2) study group (A) include 20 females with unilateral BCRL will receive kinesio taping plus manual lymphatic drainage , exercise and advices 3) study group (B) include 20 females with unilateral BCRL will receive low level laser therapy plus manual lymphatic drainage , exercise and advices 4) study group (C) include 20 females with unilateral BCRL will receive kinesio taping plus low level laser therapy and manual lymphatic drainage , exercise and advices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Experimental): study group (A) include 20 females with unilateral BCRL will receive kinesio taping plus manual lymphatic drainage , exercise and advices
  Interventions: Other: kinesio taping
- Group B (Experimental): study group (B) include 20 females with unilateral BCRL will receive low level laser therapy plus manual lymphatic drainage , exercise and advices
  Interventions: Device: Low Level Laser Therapy
- Group C (Experimental): study group (C) include 20 females with unilateral BCRL will receive kinesio taping plus low level laser therapy and manual lymphatic drainage , exercise and advices
  Interventions: Device: Low Level Laser Therapy; Other: kinesio taping

INTERVENTIONS:
Device: Low Level Laser Therapy — The device has the following treatment parametes :
  * Maximum average power > 500 milli watts
  * Wave length combined (904-808) nm
  * Maximum repition rate (1-2000) Hz
  * Energy density : 4:6 J per cm per session
  Arms: Group B; Group C
Other: kinesio taping — * the material used is 100%acrylic,latex free and heat activated with 10-15% stretch.
  * It is made of 100% cotton to allow quickening of the drying process.
  * Ability to stretch to 120-140% of its original length
  * Recoil back to the anchor that is applied without stretch
  * Heat-activated adhesive
  * Hypoallergenic dyes that make the tape safe for most users
  * Latex-free
  * Drying time after being wet is about 5-10 minutes
  * Can be worn for several days
  Arms: Group C; group A

SUMMARY:
find out the difference in the effect of kinesio taping and low level laser therapy on 66 patients with post mastectomy lymphedema as regards the following outcomes:

1.girth measurement between the upper limbs 2.) SPADI 3) hand grip strength 4)the quality of life by cancer specific questionnaire.

DETAILED DESCRIPTION:
60 females with BCRL will be recruited in this study for 4 weeks , their age ranged from 400 to 55 years old with stege 1,2 lymphedema and randomly divided into 3 equal groups: 2) study group (A) include 20 females with unilateral BCRL will receive kinesio taping plus manual lymphatic drainage , exercise and advices 3) study group (B) include 20 females with unilateral BCRL will receive low level laser therapy plus manual lymphatic drainage , exercise and advices 4) study group (C) include 20 females with unilateral BCRL will receive kinesio taping plus low level laser therapy and manual lymphatic drainage , exercise and advices regards the following outcomes:

1.girth measurement between the upper limbs 2.) SPADI 3) hand grip strength 4)the quality of life by cancer specific questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* persistence of lymphedema following mastectomy or breast conservative surgery for at least 3 months

  * minimum volume difference of 200 mL or an average difference in arm circumference of 2 cm or 10% between healthy and affected limbs.
  * Femal with unilateral lymphedema from 40 to 55 years old

Exclusion Criteria:

* • Any disease lead to swelling

  * Medication especially diuretics
  * allergy
  * infection
  * pregnancy
  * heart band kidney disease
  * bilateral lymphedema
  * skin disease
  * chronic inflammatory disease

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
girth measurment | 4 weeks
  Measurement of arm circumference is the most commonly used technique for identifying lymphedema and is reliable for both surgical and nonsurgical upper limbs It is measured using a tape with the patient in prone lying position, with elbows straight and arms relaxed at the sides. It was measured starting with 3 cm on the ulnar styloid process and proceeding with 45 cm proximal, and additionally at the metacarpal bones and mid-hand. The tape measure was put around the limb to prevent it from slacking and to ensure that there was no space in the tissue. The total circumference of the sound limb was ascertained similarly. The difference between the 2 measurements was identified using "circumference difference."
handgrip strength | 4 weeks
  evaluated using a dynamometer ,The grip strength was measured with the patient in a standing position with adducted shoulder, elbow flexed at 90°, and forearm in mid position. The patient was instructed to do 3 trials with 15 seconds rest in between each, and the highest reading was reported

SECONDARY OUTCOMES:
shoulder pain and disability index | 4 weeks
  was used to assess shoulder pain and disability. It incorporates 13 items assessing 2 domains: 5 items assess pain and 8 items evaluate disability.
quality of life questionnaire | 4 weeks
  was assessed by cancer-specific questionnaire (EORTC QLQ-C30). It is composed of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects). The functional scores ranged between 0 and 100, and higher scores indicated better condition. This questionnaire also included symptoms score (pain, dyspnea, fatigue, insomnia, nausea, loss of appetite, and financial problems). The symptom scores ranged from 100 to 0, and lower scores indicated better condition

CONTACTS AND LOCATIONS:
Overall Officials: MERIT MAGDY ZAKI, physiotherapist, Principal Investigator — beni suif university; SHERIN HASSAN MEHANI, Professor of Physical therapy, Study Chair — beni suif university; MAHMOUD AWD ELKHOLY, Lecturer of physical therapy, Study Director — beni suif university
Locations (2):
- Egypt (2):
  - Cairo University Hospital, Cairo, Cairo Governorate
  - Cairo -Beni-Suif University Hospital, GIZA, Cairo Governorate